CLINICAL TRIAL: NCT03676400
Title: Clinical Study for the Assessment of the Hair Growth Efficacy and Safety of a Cosmetic Investigational Product, After Repeated Applications for 24 Weeks, Under Normal Conditions of Use, in the Asian Adult Subjects With Androgenic Alopecia
Brief Title: Hair Growth Efficacy and Safety of NGF-574H in Adult With Androgenic Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MP-CM-001
Record Dates: First submitted 2018-09-12; First posted 2018-09-18 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Androgenic Alopecia
Keywords: mesenchymal stem cells; conditioned media; NGF-574H; hair growth; androgenic alopecia; paracrine factors; umbilical cord blood
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Product group / Control(placebo) group
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NGF-574H (Experimental): NGF-574H is hair serum with 5% conditioned media of umbilical cord blood-derived stem cells containing various trophic factors that help alleviate hair loss.
  NGF-574H will be directed to use on hair and scalp by subject her/himself at home twice a day (in the morning and evening) for 24 weeks.
  Interventions: Other: conditioned media of umbilical cord blood-derived stem cells
- placebo (Placebo Comparator): Hair serum without conditioned media of umbilical cord blood-derived stem cells will be directed to use on hair and scalp by subject her/himself at home twice a day (in the morning and evening) for 24 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: conditioned media of umbilical cord blood-derived stem cells — Hair serum with 5% conditioned media of human umbilical cord blood-derived mesenchymal stem cells
  Other Names: NGF-574H
  Arms: NGF-574H
Other: Placebo — Hair serum without conditioned media of human umbilical cord blood-derived mesenchymal stem cells
  Arms: placebo

SUMMARY:
The purpose of this study is to assess whether cosmetic investigational product containing NGF-574H is safe and effective in the treatment of androgenic alopecia in asian adults.

DETAILED DESCRIPTION:
NGF-574H is a obtained by collection of paracrine factors secreted by human umbilical cord blood-derived mesenchymal stem cell that was exposed in vitro to an artificially designed environment mimicking alopecia state in hair follicles to prime the composition of the paracrine factors optimized for hair growth. This study is to assess and confirm whether NGF-574H is safe and effective in the treatment of androgenic alopecia in asian adults.

ELIGIBILITY:
Inclusion Criteria:

1. Origin: Asian (Korean)
2. Age: adult from 18 to 60 years old
3. Sex: female (minimum 70) and male
4. Understanding of the language spoken in the research center: subjects able to read the documents they are presented with and to hold to what they are explained.
5. Social cover: subjects having medical coverage
6. Subjects whose state of health, at the moment of inclusion, (auto-questionnaires and medical examinations for the recruitment, selection and inclusion), are compatible with this type of study.
7. Subjects can be pursuit and observation during the study period.
8. Subjects have a "hair loss grade" as below criteria:

   * BASP grade: Basic type (M2 to M3, or C2 to C3, or U1 to U3) or Specific type (V1 to V3, or F1 to F3)
   * For female: Ludwig grade: Ⅰ to Ⅱ
   * For male: Norwood-Hamilton grade: III to IV
   * Hair density by phototrichogram: 60 to 190 hair/cm2
   * Telogen hair ≥ 5%
9. Subject with hair length ≥3cm in the vertex region and intending to keep this minimum length during the whole study period.
10. Subject accepting the constraints of the phototrichogram technique, i.e. agreeing to have 1 shaved zone of 1.5cm2 on the scalp.
11. Subject agreeing not to apply any topical treatment (other than the investigational product) or take any oral product or nutritional supplementation, or have any diet known to improve scalp and/or hair qualities or reduce hair loss during the whole study period.
12. Subject agreeing to use a neutral shampoo (subject's own shampoo)
13. Subject agrees to have a tattoo on the scalp on phototrichogram evaluation area.
14. Subject presenting preferably with chestnut brown, dark or black hair (in order to avoid problems of contrast)

Exclusion Criteria:

1. Subject deprived from liberty by a judiciary or administrative decision, sick subject in situation of emergency.
2. Under age or off age subject protected by law, as well as those admitted to sanitary or social facilities, ever since the research can be performed in another manner.
3. Subject who cannot be contacted in case of emergency.
4. Females in pregnancy (positive urine pregnancy-tests performed at screening(visit 1 and visit 9)or nursing or without effective contraception method.
5. Subject with any systemic disorder or skin disease (e.g. scalp disorders such as seborrheic dermatitis or scalp psoriasis) or presenting genetic or hormonal alopecia.
6. Subject with a condition or receiving a medication which, in the opinion of the investigator, could compromise the safety of the subject or affect the outcome of the study.
7. Subject using topic cosmetic treatment or oral nutritional supplement likely to interfere on hair loss parameters during the last 3 months prior to the start of the study (screening)
8. Subject having a medical treatment likely to induce an alopecia or hypertrichosia, or having stopped it from than 3 months (including prostaglandins, rubefacients agents, all vasodilators, anti-androgens, all local hormonal treatment, etc...)
9. Subject following a long period (>30 days) treatment of anti-inflammatory during the last 4 months before the start of the study (screening)
10. Subject following a short period (<30 days) treatment of anti-inflammatory stopped or ongoing preceding the screening period.
11. Subject having a immunosuppressive and/or corticoids treatment during the 4 weeks preceding the screening period
12. Subject having dyed, bleached hair or with a permanent wave prior to study start.
13. Subject who have been exposed to excessive or intensive UV light (natural or artificial) prior to the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Change in mean total hair density (hair/cm2) | 0, 6, 12 and 24 weeks
  * The hair density by phototrichogram for 24 weeks application, in comparison to initial value (baseline) and/or placebo product.
  * Measurement of hair density by phototrichogram (Canfield): change in mean total hair density (hair/cm^2)
  * Statistical analysis: Time and product effects (p<0.05)
Compare visual assessment before and after cosmetic treatment | 0, 6, 12 and 24 weeks
  Visual Assessment using the clinical picture by an investigator: 7 point score (-3 to 3) Visual assessment by a subject (Self-Assessment): 7 point score (-3 to 3)

SECONDARY OUTCOMES:
Change in mean Telogen hair density | 0, 6, 12 and 24 weeks
  Measurement of telogen hair density, in comparison to initial value (baseline) and/or placebo product.
Change in mean Anagen hair density | 0, 6, 12 and 24 weeks
  Measurement of anagen hair density, in comparison to initial value (baseline) and/or placebo product.
Change in hair growth speed | 0, 6, 12 and 24 weeks
  Measurement of hair growth speed, in comparison to initial value (baseline) and/or placebo product.
Change in hair diameter | 0, 6, 12 and 24 weeks
  Measurement of hair diameter, in comparison to initial value (baseline) and/or placebo product. Measure hair diameter using electronic outside micrometer.

CONTACTS AND LOCATIONS:
Overall Officials: Byungcheol PARK, MD, Principal Investigator — Dankook University
Locations (1):
- Dankook University Hospital, Cheonan, Chung Nam, South Korea